CLINICAL TRIAL: NCT00996567
Title: Phase II Study of Cetuximab Combined With Cisplatin or Carboplatin/Pemetrexed as First Line Treatment in Patients With Malignant Pleural Mesothelioma.
Brief Title: A Study of Cetuximab Combined With Cisplatin or Carboplatin/Pemetrexed as First Line Treatment in Patients With Malignant Pleural Mesothelioma.
Acronym: MesoMab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009/337
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Cancer
Keywords: Malignant mesothelioma
MeSH Terms: conditions — Neoplasms; Mesothelioma, Malignant | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cetuximab (Erbitux) (Experimental)
  Interventions: Drug: Cetuximab (Erbitux)

INTERVENTIONS:
Drug: Cetuximab (Erbitux) — Patients will be treated with standard chemotherapy (4-6 cycles), combined with weekly administration of Cetuximab (Erbitux) until disease progression.

SUMMARY:
Multicenter, open phase 2 study on patients with malignant mesothelioma. Standardly, 4 to 6 cycles of palliative chemotherapy, platinum in combination with pemetrexed, are given. Despite of this treatment, median survival is poor (9-12 months). By combining conventional cytotoxic agents with a novel agent, hopefully treatment and survival can be approved. Cetuximab or Erbitux is a monoclonal antibody against the EGFR (Epidermal Growth Factor Receptor). By blocking the receptor, it interferes with cel growth and division. Most mesothelioma show a strong expression of the EGFR protein. Apart from that, Cetuximab also has antibody-dependent cell-mediated cytotoxicity (ADCC).

In this trial, patients will be treated with standard chemotherapy, combined with Cetuximab weekly. After a maximum of 6 cycles of chemotherapy, administration of Cetuximab will be continued until disease progression. Every 6 weeks, a CT scan will be done to evaluate therapy. Most common side effect of Cetuximab is acneiform rash.

The translation research program consists of the determination of EGFR- and K-Ras mutations on the tumor tissue and the correlation with outcome.

In the first part of the trial, 18 patients will be included. After a positive interim analysis, a total of 43 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven malignant pleural mesothelioma, epitheloid subtype
* Recurrent after radical surgery or disease not considered suitable for radical treatment
* EGFR IHC + as assessed by DAKO kit with at least 1% of cells showing staining
* Performance status WHO 0 or 1
* Life expectancy > 12 weeks
* Weight loss < 10% in last 3 months
* Adequate bone marrow reserve, renal and hepatic function
* Measurable disease (modified RECIST)
* No prior chemotherapy
* No prior or other malignancies, except if longer than 5 yrs ago and adequately treated or basocellular skin or in situ cervical cancer
* No uncontrolled infection
* Written informed consent.
* Male/Female
* > 18 years

Exclusion Criteria:

* Evidence of brain or leptomeningeal metastases
* Patients who are unable to interrupt aspirin, other nonsteroidal anti-inflammatory drugs for a 5-day period starting 2 days before administration of pemetrexed (8-day period for long acting agents such as piroxicam)
* Patients that cannot be treated with folic acid and vitamin B 12
* Patients that cannot be treated with dexamethasone.
* Presence of clinically detectable (by physical examination) third-space fluid collections, for example ascites of pleural effusions that cannot be controlled by drainage or other procedures prior to the study entry.
* Use of investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Progression fee survival rate | At 18 weeks

SECONDARY OUTCOMES:
Response rate according to modified RECIST criteria | every 6 weeks until progression
Toxicity (CTCAE version 4) | weekly during treatment and follow-up of AE's until 30 days after last dosis
Overall survival | average survival of 9 - 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Veerle Surmont, MD, Principal Investigator — University Hospital, Ghent
Locations (4):
- Belgium (3):
  - UZ Antwerpen, Antwerp
  - University Hospital Ghent, Ghent
  - AZ St. Maarten, Mechelen
- AMC Heerlen, Heerlen, Netherlands

REFERENCES:
- See also: website of the University Hospital Ghent — http://www.uzgent.be